CLINICAL TRIAL: NCT05071352
Title: Adjuvant Continuous Infusion of Nefopam Versus Standard of Care in Mechanically Ventilated Critically Ill Patients: Randomized Double-blind Controlled Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Gamal Abdelraouf Amer, Clinical Reseacher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nefopam
Record Dates: First submitted 2021-09-04; First posted 2021-10-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2023-02

CONDITIONS: Analgesia; Critical Illness; Mechanical Ventilation; Sedation
Keywords: Nefopam, Ketamine, Standard of care, Sedation, Critically ill, Mechanical ventilation, Propofol, Fentanyl, Midazolam, Delirium, Vasopressors.
MeSH Terms: conditions — Agnosia; Critical Illness; Delirium | interventions — Nefopam; Standard of Care; Restraint, Physical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nefopam group (Experimental): Adjunct continuous infusion of nefopam plus standard of care in ICU for assessment and management of pain, sedation, and delirium.
  Nefopam will be administered as an initial dose of 20 mg IV dose infused over 15 minutes then, as continuous infusion of 5 mg/hr for 24 hours.
  Interventions: Drug: Nefopam; Drug: Standard of care in the ICU for assessment and management of pain, sedation, and delirium.
- Control group (Placebo Comparator): Standard of care in the ICU for assessment and management of pain, sedation, and delirium.
  Interventions: Drug: Standard of care in the ICU for assessment and management of pain, sedation, and delirium.

INTERVENTIONS:
Drug: Nefopam — Nefopam will be administered as an initial dose of 20 mg IV dose infused over 15 minutes then, as continuous infusion of 5 mg/hr for 24 hours.
  Other Names: Acupan
  Arms: Nefopam group
Drug: Standard of care in the ICU for assessment and management of pain, sedation, and delirium. — In our protocol we use analgiosedation approach (an opioid is used before a sedative to reach the sedation goal), targeting light sedation using richmond agitation sedation scale (RASS) score -1 to 0, and assess delirium using confusion assessment method for the ICU (CAM-ICU).
  Other Names: Standard of care

SUMMARY:
The aim of this prospective, randomized, active control, double blinded study is to assess the effect and safety of continuous infusion nefopam in mechanically ventilated ICU patients compared to standard of care. It is being hypothesized that continuous infusion nefopam will reduce opioid use with acceptable safety profile compared to standard of care.

DETAILED DESCRIPTION:
Pain is defined as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage or described in terms of such damage". Critically ill patients experience pain at rest and during standard caring procedures. Arterial catheter insertion, chest tube removal, wound drain removal, wound care, and turning are associated with the greatest increased pain intensity. Pain have short and long-term sequelae on critically ill patients. Short-term sequelae include impaired tissue oxygenation, impaired wound healing, and impaired immune functions. Long-term sequelae include chronic pain, Post-traumatic stress disorder (PTSD) symptoms, and a lower health-related quality of life.

The gold standard for pain assessment is patient's self-report of pain. For critically ill able to self-report pain the 0-10 numeric rating scale in a visual format (NRS-V) is the best to use. Unfortunately, a lot of critically ill patients are unable to communicate and self-report pain. So, using behavioral pain scales are suitable in this type of patients, Critical care pain observation tool (CPOT) demonstrates validity and reliability for monitoring pain in critical ill adult patient who are unable to self-report pain and in whom behaviors are observable. The 2018 Pain, Agitation/sedation, Delirium, Immobility, and Sleep disruption (PADIS) guideline panel suggests "using an assessment-driven, protocol-based, stepwise approach for pain and sedation management in critically ill adults" and state as a good practice statement "critically ill adults should be regularly assessed for delirium using a valid tool".

Opioids are a cornerstone in the management of pain in critically ill patient, but have a lot of negative consequences including constipation, urinary retention, bronchospasm, over-sedation, respiratory depression, hypotension, nausea, truncal rigidity, delirium, and immunosuppression. Also, they contribute to vasodilatation and hypotension which lead to increased resuscitation fluids volume in critically ill patient.

"Multi-modal analgesia" also known as "balanced analgesia" approach via using non-opioids adjuvant or in replacement of opioids to target different pain pathways leads to optimizing analgesia and reducing opioids consumption. In France, the second most prescribed non-opioids in mechanically ventilated intensive care unit (ICU) patient is nefopam. Nefopam is a non-opioid, non-steroidal centrally acting analgesic, although the exact mechanism of action poorly understood, analgesic activity is thought to be via inhibiting dopamine, norepinephrine, serotonin reuptake. Nefopam was non-inferior to fentanyl for pain control in patients undergoing elective cardiac surgery without increase in adverse effects. Nefopam has a fentanyl sparing effect up to 50% in patients underwent laparoscopic total hysterectomy.

The 2018 PADIS guideline panel made a conditional recommendation for using "nefopam (if feasible) either as an adjunct or replacement for an opioid to reduce opioid use and their safety concerns for pain management in critically ill adults".

Therefore, the aim of this prospective, randomized, active control, double blinded study is to assess the effect and safety of continuous infusion nefopam in mechanically ventilated ICU patients compared to standard of care. It is being hypothesized that continuous infusion nefopam will reduce opioid use with acceptable safety profile compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients >18 years on mechanical ventilation and expected to need ventilatory support for the next 24 hours.
2. Candidate for sedation and analgesia protocol

Exclusion Criteria:

1. Pregnant and/or lactating woman.
2. Has been intubated for duration longer than 12 hours in an intensive care unit.
3. Proven or suspected acute primary brain lesion such as traumatic brain injury, intracranial haemorrhage, stroke, or hypoxic brain injury.
4. Proven or suspected spinal cord injury or other pathology that may result in permanent or prolonged weakness.
5. Admission as a consequence of a suspected or proven drug overdose
6. Mean arterial pressure (MAP) < 50 mmHg despite adequate resuscitation and vasopressor therapy at time of randomization.
7. Death is deemed to be imminent or inevitable during this admission and either the attending physician, patient or substitute decision maker is not committed to active treatment.
8. Patients with severe hepatic impairment (Child-Pugh class C) or end stage renal disease (ESRD) (creatinine clearance < 30 ml/min or on chronic hemodialysis) due to altered pharmacokinetics [20].
9. Need for deep sedation such as administration of neuromuscular blockers.
10. Convulsions or previous history of convulsions.
11. Risk of urinary retention linked to uretroprostatic disorders.
12. Risk of acute angle glaucoma.
13. Known intolerance of or hypersensitivity to study medications or constituents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Cumulative dose of fentanyl | First 24 hour after randomization.
  To compare the cumulative dose of fentanyl

SECONDARY OUTCOMES:
Richmond Agitation and Sedation Score (RASS) | First 24 hours after randomization.
  To compare number of patients are in RASS score goal. RASS score minumum -5 (unarousable), maximun +4 (Combative). Goal RASS score from -1 (drowsy) to 0 (alert and calm).
pain score | First 24 hours after randomization.
  To compare number of patients are in Pain score goal. If patient able to communicate we use the 0-10 numeric rating scale in a visual format (NRS-V), 0 indicate no pain and 10 indicate the worst pain imaginable.
  For patient unable to communicate we use Critical care pain observation tool (CPOT) score, a score ≥3 indicate significant pain.
Duration of mechanical ventilation (MV) | The number of calendar days from intubation date to extubation date, until ICU discharge, death, or 28 days post-randomization, whichever comes first.
  To assess whether nefopam can help to shorten the of being mechanically ventilated.
vasopressor requirements | First 24 hours after randomization.
  To compare vasopressors requirement
Hemodynamics | First 24 hours after randomization.
  changes in Mean Arterial Pressure (MAP) mmHg
Hemodynamics | First 24 hours after randomization.
  changes in Heart Rate (HR) beats/minute.
ICU length of stay (LOS) | From randomization to ICU discharge date
  To compare ICU LOS
Tracheostomy | 28 days post-randomization
  Tracheostomy rate
Unplanned extubation (self-extubation) | 28 days post-randomization
  Unplanned extubation date rate
Re-intubation | 28 days post-randomization
  Re-intubation rate
Incidence of delirium | 24 hour after randomization
  Rate of positive confusion assessment method for the ICU (CAM-ICU) score
Use of antipsychotics | 24 hour after randomization
  Rate of using antipsychotics for confirmed ICU-acquired delirium
Use of physical restraint | 24 hour after randomization
  Use of physical restraint
Mortality rate at the time of hospital discharge or 28 days after randomization, whichever comes first. | 28 days after randomization
  Mortality rate at the time of hospital discharge or 28 days after randomization, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Gamal Abdelraouf Amer, Pharm D, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals (Kasr Alainy), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loeser JD, Treede RD. The Kyoto protocol of IASP Basic Pain Terminology. Pain. 2008 Jul 31;137(3):473-477. doi: 10.1016/j.pain.2008.04.025. Epub 2008 Jun 25. No abstract available. PMID 18583048
- [Background] Chanques G, Sebbane M, Barbotte E, Viel E, Eledjam JJ, Jaber S. A prospective study of pain at rest: incidence and characteristics of an unrecognized symptom in surgical and trauma versus medical intensive care unit patients. Anesthesiology. 2007 Nov;107(5):858-60. doi: 10.1097/01.anes.0000287211.98642.51. No abstract available. PMID 18073576
- [Background] Puntillo KA, Max A, Timsit JF, Vignoud L, Chanques G, Robleda G, Roche-Campo F, Mancebo J, Divatia JV, Soares M, Ionescu DC, Grintescu IM, Vasiliu IL, Maggiore SM, Rusinova K, Owczuk R, Egerod I, Papathanassoglou ED, Kyranou M, Joynt GM, Burghi G, Freebairn RC, Ho KM, Kaarlola A, Gerritsen RT, Kesecioglu J, Sulaj MM, Norrenberg M, Benoit DD, Seha MS, Hennein A, Periera FJ, Benbenishty JS, Abroug F, Aquilina A, Monte JR, An Y, Azoulay E. Determinants of procedural pain intensity in the intensive care unit. The Europain(R) study. Am J Respir Crit Care Med. 2014 Jan 1;189(1):39-47. doi: 10.1164/rccm.201306-1174OC. PMID 24262016
- [Background] Chapman CR, Tuckett RP, Song CW. Pain and stress in a systems perspective: reciprocal neural, endocrine, and immune interactions. J Pain. 2008 Feb;9(2):122-45. doi: 10.1016/j.jpain.2007.09.006. Epub 2007 Dec 21. PMID 18088561
- [Background] Tennant F. The physiologic effects of pain on the endocrine system. Pain Ther. 2013 Dec;2(2):75-86. doi: 10.1007/s40122-013-0015-x. Epub 2013 Aug 20. PMID 25135146
- [Background] Sigakis MJ, Bittner EA. Ten Myths and Misconceptions Regarding Pain Management in the ICU. Crit Care Med. 2015 Nov;43(11):2468-78. doi: 10.1097/CCM.0000000000001256. PMID 26308433
- [Background] Chanques G, Viel E, Constantin JM, Jung B, de Lattre S, Carr J, Cisse M, Lefrant JY, Jaber S. The measurement of pain in intensive care unit: comparison of 5 self-report intensity scales. Pain. 2010 Dec;151(3):711-721. doi: 10.1016/j.pain.2010.08.039. Epub 2010 Sep 16. PMID 20843604
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Gelinas C, Fillion L, Puntillo KA, Viens C, Fortier M. Validation of the critical-care pain observation tool in adult patients. Am J Crit Care. 2006 Jul;15(4):420-7. PMID 16823021
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Wibbenmeyer L, Sevier A, Liao J, Williams I, Light T, Latenser B, Lewis R 2nd, Kealey P, Rosenquist R. The impact of opioid administration on resuscitation volumes in thermally injured patients. J Burn Care Res. 2010 Jan-Feb;31(1):48-56. doi: 10.1097/BCR.0b013e3181c7ed30. PMID 20061837
- [Background] Kohler M, Chiu F, Gelber KM, Webb CA, Weyker PD. Pain management in critically ill patients: a review of multimodal treatment options. Pain Manag. 2016 Nov;6(6):591-602. doi: 10.2217/pmt-2016-0002. Epub 2016 May 18. PMID 27188977
- [Background] Kumar K, Kirksey MA, Duong S, Wu CL. A Review of Opioid-Sparing Modalities in Perioperative Pain Management: Methods to Decrease Opioid Use Postoperatively. Anesth Analg. 2017 Nov;125(5):1749-1760. doi: 10.1213/ANE.0000000000002497. PMID 29049119
- [Background] Payen JF, Genty C, Mimoz O, Mantz J, Bosson JL, Chanques G. Prescribing nonopioids in mechanically ventilated critically ill patients. J Crit Care. 2013 Aug;28(4):534.e7-12. doi: 10.1016/j.jcrc.2012.10.006. Epub 2013 Mar 19. PMID 23522398
- [Background] Gregori-Puigjane E, Setola V, Hert J, Crews BA, Irwin JJ, Lounkine E, Marnett L, Roth BL, Shoichet BK. Identifying mechanism-of-action targets for drugs and probes. Proc Natl Acad Sci U S A. 2012 Jul 10;109(28):11178-83. doi: 10.1073/pnas.1204524109. Epub 2012 Jun 18. PMID 22711801
- [Background] Kim K, Kim WJ, Choi DK, Lee YK, Choi IC, Sim JY. The analgesic efficacy and safety of nefopam in patient-controlled analgesia after cardiac surgery: A randomized, double-blind, prospective study. J Int Med Res. 2014 Jun;42(3):684-92. doi: 10.1177/0300060514525351. Epub 2014 Apr 1. PMID 24691459
- [Background] Moon JY, Choi SS, Lee SY, Lee MK, Kim JE, Lee JE, Lee SH. The Effect of Nefopam on Postoperative Fentanyl Consumption: A Randomized, Double-blind Study. Korean J Pain. 2016 Apr;29(2):110-8. doi: 10.3344/kjp.2016.29.2.110. Epub 2016 Apr 1. PMID 27103966
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Mimoz O, Chauvet S, Gregoire N, Marchand S, Le Guern ME, Saleh A, Couet W, Debaene B, Levy RH. Nefopam pharmacokinetics in patients with end-stage renal disease. Anesth Analg. 2010 Nov;111(5):1146-53. doi: 10.1213/ANE.0b013e3181f33488. PMID 20971961
- [Background] Du Manoir B, Aubrun F, Langlois M, Le Guern ME, Alquier C, Chauvin M, Fletcher D. Randomized prospective study of the analgesic effect of nefopam after orthopaedic surgery. Br J Anaesth. 2003 Dec;91(6):836-41. doi: 10.1093/bja/aeg264. PMID 14633755
- [Background] Chawla LS, Russell JA, Bagshaw SM, Shaw AD, Goldstein SL, Fink MP, Tidmarsh GF. Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3): protocol for a phase III, double-blind, randomised controlled trial. Crit Care Resusc. 2017 Mar;19(1):43-49. PMID 28215131
- [Derived] Abdelraouf MG, Farid SF, Mukhtar AM, Sabry NA. Adjuvant nefopam versus standard of care in mechanically ventilated surgical critically ill patients: A randomized, double-blind controlled study. Anaesth Crit Care Pain Med. 2025 May;44(3):101518. doi: 10.1016/j.accpm.2025.101518. Epub 2025 Apr 16. PMID 40250620